CLINICAL TRIAL: NCT04964063
Title: A Real-World Evidence Study Evaluating Oral Health Related Quality of Life Following the Use of Antisensitivity Toothpaste for Dentine Hypersensitivity Management
Brief Title: A Real-World Evidence Study to Evaluate Oral Health Related Quality of Life Using an Anti-Sensitivity Toothpaste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 216953
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Results first posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-04

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Sensodyne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sensodyne Fresh Mint Toothpaste (Other): Participants will be asked to follow commercial tube instructions as recommended for sensitivity relief: "Apply at least a 1-inch strip of the product onto a soft bristle toothbrush. Brush teeth thoroughly for at least 1 minute twice a day (morning and evening), and not more than 3 times a day, or as recommended by a dentist or doctor. Make sure to brush all sensitive areas of the teeth. Minimize swallowing, Spit out after brushing."
  Interventions: Other: Potassium Nitrate + Sodium Fluoride

INTERVENTIONS:
Other: Potassium Nitrate + Sodium Fluoride — Potassium Nitrate 5% weight/weight (w/w) and Sodium Fluoride 0.15% weight/volume (w/v) fluoride ion.

SUMMARY:
The purpose of this study is to evaluate changes in oral health-related quality of life (OHrQoL) in participants suffering from Dentinal Hypersensitivity (DH) symptoms following the use of anti-sensitivity toothpaste for 24 weeks.

DETAILED DESCRIPTION:
This study will be a virtual, prospective, twenty-four weeks, open label study in participants with DH (self-reported symptoms). Participants self-perception of DH will be evaluated by completion of a validated OHrQoL questionnaire (Dentin Hypersensitivity Experience Questionnaire-48 [DHEQ-48]) at baseline, 4, 8, 12, 16, 20 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of consent indicating that the participant has been informed of all pertinent aspects of the study.
* The participant must be able to complete all activities as shown in the Schedule of Activities independently on their smart devices.
* Participant who has tooth sensitivity (self-reported symptoms).

Exclusion Criteria:

* A participant whose sensitivity could be caused by other factors or clinical pathology as established by the screening questionnaire, which also includes:

  * A participant who has been/is on multiple prescription medications to treat severe acid reflux on regular basis or considered surgery for acid reflux
  * A participant with full or partial denture
  * A participant who has undergone treatment within 6 months of screening or is currently under treatment for periodontal or gum disease
  * A participant with active periodontitis
  * A participant with active caries
  * A participant with any chronic and/or severe painful health conditions which lead to regular use pain medications (more than 3 days a week)
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients: potassium nitrate (5 percent [%]), sodium fluoride (0.15% weight/volume [w/v] fluoride ion), water, sorbitol, hydrated silica, glycerin, cocamidopropyl betaine, flavor, xanthan gum, titanium dioxide, sodium saccharin, sodium hydroxide, sucralose, yellow 10, blue 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 655 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — OBVIO HEALTH USA, Inc.
Locations (1):
- GSK Investigational Site, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a decentralized, prospective, 24-weeks, open label study in participants with dentine hypersensitivity (DH) (self-reported symptoms). All the participants were recruited through social media and other digital platforms.
Pre-assignment Details: A total of 801 participants were screened, 655 were enrolled, and 557 completed the study. A total of 98 participants discontinued the study.
Groups:
- Sensodyne Fresh Mint Toothpaste: Participants were asked to follow commercial tube instructions as recommended for sensitivity relief. Participants applied dentifrice containing 5 percent (%) weight/weight (w/w) potassium nitrate and 0.15% weight/volume (w/v) sodium fluoride oral topically for 24 weeks.
Period: Overall Study
Arm/Group | Sensodyne Fresh Mint Toothpaste
Started | 655
Completed | 557
Not Completed | 98
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 47
Not completed — Withdrawal by Subject | 5
Not completed — Baseline Tasks Expired | 41
Not completed — Participant withdrawn in error | 1

BASELINE CHARACTERISTICS:
Population: The modified Intent-To-Treat (mITT) population included all participants who had received at least one dose of study product and have at least one post baseline Dentine Hypersensitivity Experience Questionnaire (DHEQ)-48 questionnaire data.
Groups:
- Sensodyne Fresh Mint Toothpaste: Participants were asked to follow commercial tube instructions as recommended for sensitivity relief. Participants applied dentifrice containing 5% w/w potassium nitrate and 0.15% w/v sodium fluoride oral topically for 24 weeks.
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 577
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.84 (10.875)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 446
  Male | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 86
  Not Hispanic or Latino | 483
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 63
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 118
  White | 353
  More than one race | 13
  Unknown or Not Reported | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Score of DHEQ Section 1 - Impact on Everyday Life (Question [Q]1-3) at Baseline (Day 0)
Description: All the participants scored question No. 1 to 3 ([Q1: On a scale of 1 to 10 how intense were the sensations?] of section 1 of DHEQ on a scale of 1 to 10, where 1 is equal to (=) not at all intense and 10= worst imaginable, [Q2: On a scale of 1 to 10 how bothered were you by any sensations?] of section 1 of DHEQ on a scale of 1 to 10, where 1= Not at all bothered and 10= Extremely bothered], [Q3: On a scale of 1 to 10 how well could you tolerate sensations?] of section 1 of DHEQ on a scale of 1 to 10, where 1= Can easily tolerate and 10= Can't tolerate at all]). Section 1 of DHEQ consisted of questions about participant's sensitive teeth and the impact they had on participant's everyday life. Lower is the score, better is the improvement in Oral Health-related Quality of Life (OHrQoL). Baseline was defined as Day 0 value.
Time Frame: Baseline (Day 0)
Population: mITT Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 577
score on a scale
  Q1: How intense are the sensation | 5.90 (1.731)
  Q2: How bothered are you by any sensation | 6.17 (2.045)
  Q3: How well can you tolerate sensations | 5.20 (2.088)

2. Primary Outcome: Mean Score of DHEQ Section 1 - Impact on Everyday Life (Q1-3) at Week 4
Description: All the participants scored question No. 1 to 3 ([Q1: On a scale of 1 to 10 how intense were the sensations?] of section 1 of DHEQ on a scale of 1 to 10, where 1= not at all intense and 10= worst imaginable, [Q2: On a scale of 1 to 10 how bothered were you by any sensations?] of section 1 of DHEQ on a scale of 1 to 10, where 1= Not at all bothered and 10= Extremely bothered], [Q3: On a scale of 1 to 10 how well could you tolerate sensations?] of section 1 of DHEQ on a scale of 1 to 10, where 1= Can easily tolerate and 10= Can't tolerate at all]). Section 1 of DHEQ consisted of questions about participant's sensitive teeth and the impact they had on participant's everyday life. Lower is the score, better is the improvement in OHrQoL.
Time Frame: Week 4
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 546
Score on a scale
  Q1: How intense are the sensation | 4.54 (1.949)
  Q2: How bothered are you by any sensation | 4.51 (2.149)
  Q3: How well can you tolerate sensations | 3.98 (2.095)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -1.33, 95% CI 2-sided [-1.47 to -1.19], Standard Error of Mean 0.08 — Q1: How intense are the sensation
Statistical Analysis 2: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -1.61, 95% CI 2-sided [-1.77 to -1.45], Standard Error of Mean 0.09 — Q2: How bothered are you by any sensation
Statistical Analysis 3: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -1.17, 95% CI 2-sided [-1.33 to -1.00], Standard Error of Mean 0.09 — Q3: How well can you tolerate sensations

3. Primary Outcome: Mean Score of DHEQ Section 1 - Impact on Everyday Life (Q1-3) at Week 8
Description: All the participants scored question No. 1 to 3 ([Q1: On a scale of 1 to 10 how intense are the sensations?] of section 1 of DHEQ on a scale of 1 to 10, where 1= not at all intense and 10= worst imaginable, [Q2: On a scale of 1 to 10 how bothered are you by any sensations?] of section 1 of DHEQ on a scale of 1 to 10, where 1= Not at all bothered and 10= Extremely bothered], [Q3: On a scale of 1 to 10 how well can you tolerate sensations?] of section 1 of DHEQ on a scale of 1 to 10, where 1= Can easily tolerate and 10= Can't tolerate at all]). Section 1 of DHEQ consisted of questions about participant's sensitive teeth and the impact they had on participant's everyday life. Lower is the score, better is the improvement in OHrQoL.
Time Frame: Week 8
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 570
Score on a scale
  Q1: How intense are the sensation | 4.06 (1.924)
  Q2: How bothered are you by any sensation | 3.99 (2.183)
  Q3: How well can you tolerate sensations | 3.74 (2.140)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Median Difference (Final Values) = -1.84, 95% CI 2-sided [-1.98 to -1.70], Standard Error of Mean 0.08 — Q1: How intense are the sensation
Statistical Analysis 2: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -2.17, 95% CI 2-sided [-2.33 to -2.02], Standard Error of Mean 0.09 — Q2: How bothered are you by any sensation
Statistical Analysis 3: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -1.45, 95% CI 2-sided [-1.61 to -1.29], Standard Error of Mean 0.09 — Q3: How well can you tolerate sensations

4. Primary Outcome: Mean Score of DHEQ Section 1 - Impact on Everyday Life (Q1-3) at Week 12
Description: as for outcome 3
Time Frame: Week 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 564
Score on a scale
  Q1: How intense are the sensation | 3.61 (1.835)
  Q2: How bothered are you by any sensation | 3.55 (2.007)
  Q3: How well can you tolerate sensations | 3.33 (1.949)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -2.29, 95% CI 2-sided [-2.43 to -2.15], Standard Error of Mean 0.08 — Q1: How intense are the sensation
Statistical Analysis 2: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -2.63, 95% CI 2-sided [-2.79 to -2.47], Standard Error of Mean 0.09 — Q2: How bothered are you by any sensation
Statistical Analysis 3: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -1.86, 95% CI 2-sided [-2.02 to -1.70], Standard Error of Mean 0.09 — Q3: How well can you tolerate sensations

5. Primary Outcome: Mean Score of DHEQ Section 1 - Impact on Everyday Life (Q1-3) at Week 16
Description: as for outcome 3
Time Frame: Week 16
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 549
Score on a scale
  Q1: How intense are the sensation | 3.34 (1.892)
  Q2: How bothered are you by any sensation | 3.26 (1.978)
  Q3: How well can you tolerate sensations | 3.14 (2.018)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -2.54, 95% CI 2-sided [-2.68 to -2.40], Standard Error of Mean 0.08 — Q1: How intense are the sensation
Statistical Analysis 2: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -2.89, 95% CI 2-sided [-3.05 to -2.73], Standard Error of Mean 0.09 — Q2: How bothered are you by any sensation
Statistical Analysis 3: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -2.04, 95% CI 2-sided [-2.20 to -1.87], Standard Error of Mean 0.09 — Q3: How well can you tolerate sensations

6. Primary Outcome: Mean Score of DHEQ Section 1 - Impact on Everyday Life (Q1-3) at Week 20
Description: as for outcome 3
Time Frame: Week 20
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 522
Score on a scale
  Q1: How intense are the sensation | 3.20 (1.959)
  Q2: How bothered are you by any sensation | 3.18 (2.041)
  Q3: How well can you tolerate sensations | 3.02 (2.015)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -2.69, 95% CI 2-sided [-2.84 to -2.55], Standard Error of Mean 0.08 — Q1: How intense are the sensation
Statistical Analysis 2: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -2.99, 95% CI 2-sided [-3.15 to -2.83], Standard Error of Mean 0.09 — Q2: How bothered are you by any sensation
Statistical Analysis 3: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -2.18, 95% CI 2-sided [-2.35 to -2.02], Standard Error of Mean 0.09 — Q3: How well can you tolerate sensations

7. Primary Outcome: Mean Score of DHEQ Section 1 - Impact on Everyday Life (Q1-3) at Week 24
Description: as for outcome 3
Time Frame: Week 24
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 560
Score on a scale
  Q1: How intense are the sensation | 2.96 (1.861)
  Q2: How bothered are you by any sensation | 2.93 (1.969)
  Q3: How well can you tolerate sensations | 2.81 (1.957)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Median Difference (Final Values) = -2.94, 95% CI 2-sided [-3.08 to -2.79], Standard Error of Mean 0.08 — Q1: How intense are the sensation
Statistical Analysis 2: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Median Difference (Final Values) = -3.24, 95% CI 2-sided [-3.40 to -3.08], Standard Error of Mean 0.09 — Q2: How bothered are you by any sensation
Statistical Analysis 3: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -2.37, 95% CI 2-sided [-2.53 to -2.21], Standard Error of Mean 0.09 — Q3: How well can you tolerate sensations

8. Primary Outcome: Mean Score of DHEQ Section 2 - Total Score (Q1-34) at Baseline (Day 0)
Description: All participants scored 34 questions present in section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6= Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Section 2 included questions assessing how sensitivity impacts the way a participant acts and feels. Total score was derived from the sum of scores of all 34 questions present in section 2 of the DHEQ. Total scores range from 238 to 34 points, lower is the score, better is the improvement in OHrQoL. Baseline was defined as Day 0 value.
Time Frame: Baseline (Day 0)
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 577
Score on a scale | 165.20 (35.554)

9. Primary Outcome: Mean Score of DHEQ Section 2 - Total Score (Q1-34) at Week 4
Description: All participants scored 34 questions present in section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6= Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Section 2 included questions assessing how sensitivity impacts the way a participant acts and feels. Total score was derived from the sum of scores of all 34 questions present in section 2 of the DHEQ. Total scores range from 238 to 34 points, lower is the score, better is the improvement in OHrQoL.
Time Frame: Week 4
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 546
Score on a scale | 145.31 (39.881)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -17.93, 95% CI 2-sided [-20.81 to -15.05], Standard Error of Mean 1.91

10. Primary Outcome: Mean Score of DHEQ Section 2 - Total Score (Q1-34) at Week 8
Description: as for outcome 9
Time Frame: Week 8
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 570
Score on a scale | 133.93 (45.319)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -31.20, 95% CI 2-sided [-34.04 to -28.36], Standard Error of Mean 1.90

11. Primary Outcome: Mean Score of DHEQ Section 2 - Total Score (Q1-34) at Week 12
Description: as for outcome 9
Time Frame: Week 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 564
Score on a scale | 125.41 (47.315)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -39.45, 95% CI 2-sided [-42.30 to -36.59], Standard Error of Mean 1.90

12. Primary Outcome: Mean Score of DHEQ Section 2 - Total Score (Q1-34) at Week 16
Description: as for outcome 9
Time Frame: Week 16
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 549
Score on a scale | 120.48 (49.014)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -44.37, 95% CI 2-sided [-47.24 to -41.49], Standard Error of Mean 1.91

13. Primary Outcome: Mean Score of DHEQ Section 2 - Total Score (Q1-34) at Week 20
Description: as for outcome 9
Time Frame: Week 20
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 522
Score on a scale | 116.98 (50.437)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -48.04, 95% CI 2-sided [-50.96 to -45.12], Standard Error of Mean 1.93

14. Primary Outcome: Mean Score of DHEQ Section 2 - Total Score (Q1-34) at Week 24
Description: as for outcome 9
Time Frame: Week 24
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 560
Score on a scale | 112.62 (50.250)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -52.47, 95% CI 2-sided [-55.33 to -49.62], Standard Error of Mean 1.91

15. Primary Outcome: Mean Score of DHEQ Section 2 - Restrictions (Q1-4) at Baseline (Day 0)
Description: All participants scored 4 questions present in Domain "Restriction" of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6= Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Restriction domain consisted of questions Q1-Q4. Domain Restriction score was derived by sum of Q1-Q4 (section 2 DHEQ). Domain Restriction scores range from 28-4, lower is the score, better is the improvement in OHrQoL. Baseline was defined as Day 0 value.
Time Frame: Baseline (Day 0)
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 577
Score on a scale | 21.56 (4.417)

16. Primary Outcome: Mean Score of DHEQ Section 2 - Restrictions (Q1-4) at Week 4
Description: All participants scored 4 questions present in Domain "Restriction" of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6= Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Restriction domain consisted of questions Q1-Q4. Domain Restriction score was derived by sum of Q1-Q4 (section 2 DHEQ). Domain Restriction scores range from 28-4, lower is the score, better is the improvement in OHrQoL.
Time Frame: Week 4
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 546
Score on a scale | 18.92 (5.432)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -2.45, 95% CI 2-sided [-2.88 to -2.02], Standard Error of Mean 0.26

17. Primary Outcome: Mean Score of DHEQ Section 2 - Restrictions (Q1-4) at Week 8
Description: as for outcome 16
Time Frame: Week 8
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 570
Score on a scale | 17.28 (6.068)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -4.27, 95% CI 2-sided [-4.69 to -3.85], Standard Error of Mean 0.25

18. Primary Outcome: Mean Score of DHEQ Section 2 - Restrictions (Q1-4) at Week 12
Description: as for outcome 16
Time Frame: Week 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 564
Score on a scale | 15.80 (6.344)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -5.71, 95% CI 2-sided [-6.13 to -5.28], Standard Error of Mean 0.25

19. Primary Outcome: Mean Score of DHEQ Section 2 - Restrictions (Q1-4) at Week 16
Description: as for outcome 16
Time Frame: Week 16
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 549
Score on a scale | 15.04 (6.512)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -6.45, 95% CI 2-sided [-6.88 to -6.02], Standard Error of Mean 0.26

20. Primary Outcome: Mean Score of DHEQ Section 2 - Restrictions (Q1-4) at Week 20
Description: as for outcome 16
Time Frame: Week 20
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 522
Score on a scale | 14.52 (6.724)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Median Difference (Final Values) = -7.01, 95% CI 2-sided [-7.45 to -6.58], Standard Error of Mean 0.26

21. Primary Outcome: Mean Score of DHEQ Section 2 - Restrictions (Q1-4) at Week 24
Description: as for outcome 16
Time Frame: Week 24
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 560
Score on a scale | 14.11 (6.774)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -7.44, 95% CI 2-sided [-7.87 to -7.01], Standard Error of Mean 0.25

22. Primary Outcome: Mean Score of DHEQ Section 2 - Adaptation (Q5-16) at Baseline (Day 0)
Description: All participants scored 12 questions present in Domain "Adaptation" of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6=Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Adaptation domain consisted of 12 questions (Q5-16). Adaptation domain score was derived by sum of Q5-Q16 (section 2 DHEQ). Domain Adaptation scores range from 84-12, lower is the score, better is the improvement in OHrQoL. Baseline was defined as Day 0 value.
Time Frame: Baseline (Day 0)
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 577
Score on a scale | 59.33 (13.761)

23. Primary Outcome: Mean Score of DHEQ Section 2 - Adaptation (Q5-16) at Week 4
Description: All participants scored 12 questions present in Domain "Adaptation" of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6=Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Adaptation domain consisted of 12 questions (Q5-16). Adaptation domain score was derived by sum of Q5-Q16 (section 2 DHEQ). Domain Adaptation scores range from 84-12, lower is the score, better is the improvement in OHrQoL.
Time Frame: Week 4
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 546
Score on a scale | 52.34 (15.206)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -6.33, 95% CI 2-sided [-7.46 to -5.20], Standard Error of Mean 0.72

24. Primary Outcome: Mean Score of DHEQ Section 2 - Adaptation (Q5-16) at Week 8
Description: as for outcome 23
Time Frame: Week 8
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 570
Score on a scale | 47.80 (17.266)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -11.53, 95% CI 2-sided [-12.64 to -10.41], Standard Error of Mean 0.72

25. Primary Outcome: Mean Score of DHEQ Section 2 - Adaptation (Q5-16) at Week 12
Description: as for outcome 23
Time Frame: Week 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 564
Score on a scale | 44.71 (17.749)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -14.54, 95% CI 2-sided [-15.66 to -13.42], Standard Error of Mean 0.72

26. Primary Outcome: Mean Score of DHEQ Section 2 - Adaptation (Q5-16) at Week 16
Description: as for outcome 23
Time Frame: Week 16
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 549
Score on a scale | 42.71 (18.378)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Median Difference (Final Values) = -16.54, 95% CI 2-sided [-17.67 to -15.41], Standard Error of Mean 0.72

27. Primary Outcome: Mean Score of DHEQ Section 2 - Adaptation (Q5-16) at Week 20
Description: as for outcome 23
Time Frame: Week 20
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 522
Score on a scale | 41.59 (18.911)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -17.73, 95% CI 2-sided [-18.87 to -16.58], Standard Error of Mean 0.73

28. Primary Outcome: Mean Score of DHEQ Section 2 - Adaptation (Q5-16) at Week 24
Description: as for outcome 23
Time Frame: Week 24
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 560
Score on a scale | 40.48 (18.578)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -18.84, 95% CI 2-sided [-19.96 to -17.72], Standard Error of Mean 0.72

29. Primary Outcome: Mean Score of DHEQ Section 2 - Social Impact (Q17-21) at Baseline (Day 0)
Description: All participants scored 5 questions present in Domain "Social Impact" of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6= Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Social Impact domain consisted of questions Q17-Q21. Social Impact domain score was derived by sum of Q17-Q21 (section 2 DHEQ). Scores range from 35-5, lower is the score, better is the improvement in OHrQoL. Baseline was defined as Day 0 value.
Time Frame: Baseline (Day 0)
Population: mITT population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 577
Score on a scale | 21.35 (6.847)

30. Primary Outcome: Mean Score of DHEQ Section 2 - Social Impact (Q17-21) at Week 4
Description: All participants scored 5 questions present in Domain "Social Impact" of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6= Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Social Impact domain consisted of questions Q17-Q21. Social Impact domain score was derived by sum of Q17-Q21 (section 2 DHEQ). Scores range from 35-5, lower is the score, better is the improvement in OHrQoL.
Time Frame: Week 4
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 546
Score on a scale | 18.95 (7.026)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -2.04, 95% CI 2-sided [-2.52 to -1.56], Standard Error of Mean 0.31

31. Primary Outcome: Mean Score of DHEQ Section 2 - Social Impact (Q17-21) at Week 8
Description: as for outcome 30
Time Frame: Week 8
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 570
Score on a scale | 17.64 (7.531)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -3.69, 95% CI 2-sided [-4.17 to -3.22], Standard Error of Mean 0.31

32. Primary Outcome: Mean Score of DHEQ Section 2 - Social Impact (Q17-21) at Week 12
Description: as for outcome 30
Time Frame: Week 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 564
Score on a scale | 16.61 (7.708)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -4.67, 95% CI 2-sided [-5.15 to -4.20], Standard Error of Mean 0.31

33. Primary Outcome: Mean Score of DHEQ Section 2 - Social Impact (Q17-21) at Week 16
Description: as for outcome 30
Time Frame: Week 16
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 549
Score on a scale | 16.06 (7.713)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -5.24, 95% CI 2-sided [-5.72 to -4.76], Standard Error of Mean 0.31

34. Primary Outcome: Mean Score of DHEQ Section 2 - Social Impact (Q17-21) at Week 20
Description: as for outcome 30
Time Frame: Week 20
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 522
Score on a scale | 15.68 (7.785)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -5.63, 95% CI 2-sided [-6.12 to -5.14], Standard Error of Mean 0.32

35. Primary Outcome: Mean Score of DHEQ Section 2 - Social Impact (Q17-21) at Week 24
Description: as for outcome 30
Time Frame: Week 24
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 560
Score on a scale | 15.08 (7.722)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -6.24, 95% CI 2-sided [-6.72 to -5.77], Standard Error of Mean 0.31

36. Primary Outcome: Mean Score of DHEQ Section 2 - Emotional Impact (Q22-29) at Baseline (Day 0)
Description: All participants scored 8 questions present in Domain "Emotional Impact" of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6=Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Emotional Impact domain consisted of questions Q22- Q29. Emotional Impact domain score was derived by sum of Q22-Q29 (section 2 DHEQ). Scores range from 56-8, lower is the score, better is the improvement in OHrQoL. Baseline was defined as Day 0 value.
Time Frame: Baseline (Day 0)
Population: mITT population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 577
Score on a scale | 41.10 (8.279)

37. Primary Outcome: Mean Score of DHEQ Section 2 - Emotional Impact (Q22-29) at Week 4
Description: All participants scored 8 questions present in Domain "Emotional Impact" of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6=Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Emotional Impact domain consisted of questions Q22- Q29. Emotional Impact domain score was derived by sum of Q22-Q29 (section 2 DHEQ). Scores range from 56-8, lower is the score, better is the improvement in OHrQoL.
Time Frame: Week 4
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 546
Score on a scale | 35.42 (10.132)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -5.25, 95% CI 2-sided [-6.06 to -4.44], Standard Error of Mean 0.48

38. Primary Outcome: Mean Score of DHEQ Section 2 - Emotional Impact (Q22-29) at Week 8
Description: as for outcome 37
Time Frame: Week 8
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 570
Score on a scale | 32.55 (11.197)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -8.52, 95% CI 2-sided [-9.32 to -7.72], Standard Error of Mean 0.47

39. Primary Outcome: Mean Score of DHEQ Section 2 - Emotional Impact (Q22-29) at Week 12
Description: as for outcome 37
Time Frame: Week 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 564
Score on a scale | 30.48 (11.959)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -10.55, 95% CI 2-sided [-11.35 to -9.75], Standard Error of Mean 0.48

40. Primary Outcome: Mean Score of DHEQ Section 2 - Emotional Impact (Q22-29) at Week 16
Description: as for outcome 37
Time Frame: Week 16
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 549
Score on a scale | 29.43 (12.425)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -11.60, 95% CI 2-sided [-12.41 to -10.79], Standard Error of Mean 0.48

41. Primary Outcome: Mean Score of DHEQ Section 2 - Emotional Impact (Q22-29) at Week 20
Description: as for outcome 37
Time Frame: Week 20
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 522
Score on a scale | 28.42 (12.630)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -12.63, 95% CI 2-sided [-13.45 to -11.81], Standard Error of Mean 0.48

42. Primary Outcome: Mean Score of DHEQ Section 2 - Emotional Impact (Q22-29) at Week 24
Description: as for outcome 37
Time Frame: Week 24
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 560
Score on a scale | 27.18 (12.641)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -13.88, 95% CI 2-sided [-14.69 to -13.08], Standard Error of Mean 0.48

43. Primary Outcome: Mean Score of DHEQ Section 2 - Identity (Q30-34) at Baseline (Day 0)
Description: All participants scored 5 questions present in Domain "Identity" of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6= Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Identity domain consisted of questions Q30- Q34. Identity domain score was derived by sum of Q30-34 (section 2 DHEQ). Scores range from 35-5, lower is the score, better is the improvement in OHrQoL. Baseline was defined as Day 0 value.
Time Frame: Baseline (Day 0)
Population: mITT population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 577
Score on a scale | 21.86 (7.800)

44. Primary Outcome: Mean Score of DHEQ Section 2 - Identity (Q30-34) at Week 4
Description: All participants scored 5 questions present in Domain "Identity" of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6= Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Identity domain consisted of questions Q30- Q34. Identity domain score was derived by sum of Q30-34 (section 2 DHEQ). Scores range from 35-5, lower is the score, better is the improvement in OHrQoL.
Time Frame: Week 4
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 546
Score on a scale | 19.68 (7.847)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -1.88, 95% CI 2-sided [-2.43 to -1.33], Standard Error of Mean 0.35

45. Primary Outcome: Mean Score of DHEQ Section 2 - Identity (Q30-34) at Week 8
Description: as for outcome 44
Time Frame: Week 8
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 570
Score on a scale | 18.66 (8.402)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -3.20, 95% CI 2-sided [-3.74 to -2.65], Standard Error of Mean 0.35

46. Primary Outcome: Mean Score of DHEQ Section 2 - Identity (Q30-34) at Week 12
Description: as for outcome 44
Time Frame: Week 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 564
Score on a scale | 17.82 (8.573)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -3.98, 95% CI 2-sided [-4.53 to -3.44], Standard Error of Mean 0.35

47. Primary Outcome: Mean Score of DHEQ Section 2 - Identity (Q30-34) at Week 16
Description: as for outcome 44
Time Frame: Week 16
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 549
Score on a scale | 17.24 (8.754)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -4.55, 95% CI 2-sided [-5.10 to -4.00], Standard Error of Mean 0.35

48. Primary Outcome: Mean Score of DHEQ Section 2 - Identity (Q30-34) at Week 20
Description: as for outcome 44
Time Frame: Week 20
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 522
Score on a scale | 16.76 (8.708)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Median Difference (Final Values) = -5.04, 95% CI 2-sided [-5.60 to -4.48], Standard Error of Mean 0.36

49. Primary Outcome: Mean Score of DHEQ Section 2 - Identity (Q30-34) at Week 24
Description: as for outcome 44
Time Frame: Week 24
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 560
Score on a scale | 15.78 (8.765)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -6.07, 95% CI 2-sided [-6.62 to -5.53], Standard Error of Mean 0.35

50. Primary Outcome: Mean Score of DHEQ Section 2 - Global Oral Health Score (Q35) at Baseline (Day 0)
Description: All participants scored one question (Q35) of section 2 of DHEQ to asses Domain "Global oral health" using 6-point scale, where 6=Very poor, 5= poor, 4= Fair, 3= Good, 2= Very good, and 1= excellent. Global oral health domain consisted of Q35. Scores range from 6-1, lower is the score, better is the improvement in OHrQoL. Baseline was defined as Day 0 value.
Time Frame: Baseline (Day 0)
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 577
Score on a scale | 2.90 (0.935)

51. Primary Outcome: Mean Score of DHEQ Section 2 - Global Oral Health Score (Q35) at Week 4
Description: All participants scored one question (Q35) of section 2 of DHEQ to asses Domain "Global oral health" using 6-point scale, where 6=Very poor, 5= poor, 4= Fair, 3= Good, 2= Very good, and 1= excellent. Global oral health domain consisted of Q35. Scores range from 6-1, lower is the score, better is the improvement in OHrQoL.
Time Frame: Week 4
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 546
Score on a scale | 2.83 (0.887)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p = 0.1091, ANOVA; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.12 to 0.01], Standard Error of Mean 0.04

52. Primary Outcome: Mean Score of DHEQ Section 2 - Global Oral Health Score (Q35) at Week 8
Description: as for outcome 51
Time Frame: Week 8
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 570
Score on a scale | 2.78 (0.883)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.19 to -0.06], Standard Error of Mean 0.04

53. Primary Outcome: Mean Score of DHEQ Section 2 - Global Oral Health Score (Q35) at Week 12
Description: as for outcome 51
Time Frame: Week 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 564
Score on a scale | 2.74 (0.906)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.23 to -0.10], Standard Error of Mean 0.04

54. Primary Outcome: Mean Score of DHEQ Section 2 - Global Oral Health Score (Q35) at Week 16
Description: as for outcome 51
Time Frame: Week 16
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 549
Score on a scale | 2.72 (0.904)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.24 to -0.11], Standard Error of Mean 0.04

55. Primary Outcome: Mean Score of DHEQ Section 2 - Global Oral Health Score (Q35) at Week 20
Description: as for outcome 51
Time Frame: Week 20
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 522
Score on a scale | 2.69 (0.917)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Median Difference (Final Values) = -0.19, 95% CI 2-sided [-0.26 to -0.13], Standard Error of Mean 0.04

56. Primary Outcome: Mean Score of DHEQ Section 2 - Global Oral Health Score (Q35) at Week 24
Description: as for outcome 51
Time Frame: Week 24
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 560
Score on a scale | 2.65 (0.898)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.31 to -0.18], Standard Error of Mean 0.04

57. Primary Outcome: Mean Score of DHEQ Section 2 - Effect of Life Overall Score (Q36 - 39) at Baseline (Day 0)
Description: All participants scored 4 questions present in Domain "Effect on Life Overall" of section 2 of the DHEQ using a 5-point scale, 4= Very Much, 3= Quite a bit, 2= somewhat, and 1= a little, 0=not at all. Effect on Life Overall domain consisted of Q36 - 39. Effect on Life Overall domain score was derived by sum of Q36-39 (section 2 DHEQ). Scores range from 20-0, lower is the score, better is the improvement in OHrQoL. Baseline was defined as Day 0 value.
Time Frame: Baseline (Day 0)
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 577
Score on a scale | 8.52 (3.326)

58. Primary Outcome: Mean Score of DHEQ Section 2 - Effect of Life Overall Score (Q36 - 39) at Week 4
Description: All participants scored 4 questions present in Domain "Effect on Life Overall" of section 2 of the DHEQ using a 5-point scale, 4= Very Much, 3= Quite a bit, 2= somewhat, and 1= a little, 0=not at all. Effect on Life Overall domain consisted of Q36 - 39. Effect on Life Overall domain score was derived by sum of Q36-39 (section 2 DHEQ). Scores range from 20-0, lower is the score, better is the improvement in OHrQoL.
Time Frame: Week 4
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 546
Score on a scale | 6.71 (3.190)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -1.70, 95% CI 2-sided [-1.95 to -1.45], Standard Error of Mean 0.14

59. Primary Outcome: Mean Score of DHEQ Section 2 - Effect of Life Overall Score (Q36 - 39) at Week 8
Description: as for outcome 58
Time Frame: Week 8
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 570
Score on a scale | 5.81 (3.304)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -2.69, 95% CI 2-sided [-2.94 to -2.44], Standard Error of Mean 0.14

60. Primary Outcome: Mean Score of DHEQ Section 2 - Effect of Life Overall Score (Q36 - 39) at Week 12
Description: as for outcome 58
Time Frame: Week 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 564
Score on a scale | 5.41 (3.410)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -3.09, 95% CI 2-sided [-3.35 to -2.84], Standard Error of Mean 0.14

61. Primary Outcome: Mean Score of DHEQ Section 2 - Effect of Life Overall Score (Q36 - 39) at Week 16
Description: as for outcome 58
Time Frame: Week 16
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 549
Score on a scale | 5.05 (3.404)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -3.44, 95% CI 2-sided [-3.69 to -3.19], Standard Error of Mean 0.14

62. Primary Outcome: Mean Score of DHEQ Section 2 - Effect of Life Overall Score (Q36 - 39) at Week 20
Description: as for outcome 58
Time Frame: Week 20
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 522
Score on a scale | 4.69 (3.362)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Median Difference (Final Values) = -3.80, 95% CI 2-sided [-4.06 to -3.55], Standard Error of Mean 0.14

63. Primary Outcome: Mean Score of DHEQ Section 2 - Effect of Life Overall Score (Q36 - 39) at Week 24
Description: as for outcome 58
Time Frame: Week 24
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sensodyne Fresh Mint Toothpaste
Number analyzed (Participants) | 560
Score on a scale | 4.25 (3.421)
Statistical Analysis 1: Comparison: Sensodyne Fresh Mint Toothpaste; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -4.26, 95% CI 2-sided [-4.51 to -4.00], Standard Error of Mean 0.14

ADVERSE EVENTS:
Time Frame: From screening up to Week 24, up to approximately 168 days
Description: An Adverse Event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product (or medical device). A Serious Adverse Event (SAE) is a particular category of an adverse event where the adverse outcome is serious.
Arm/Group | Sensodyne Fresh Mint Toothpaste
All-Cause Mortality (participants affected / at risk) | 0/584
Serious Adverse Events (participants affected / at risk) | 2/584
Other Adverse Events (participants affected / at risk) | 41/584
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensodyne Fresh Mint Toothpaste (N=584)
Head Injury (Injury, poisoning and procedural complications) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sensodyne Fresh Mint Toothpaste (N=584)
Covid-19 (Infections and infestations) | 11
Nasopharyngitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Pharyngitis Streptococcal (Infections and infestations) | 1
Attention Deficit Hyperactivity Disorder (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Post-Traumatic Stress Disorder (Psychiatric disorders) | 2
Borderline Personality Disorder (Psychiatric disorders) | 1
Hallucination, Auditory (Psychiatric disorders) | 1
Hallucination, Visual (Psychiatric disorders) | 1
Cheilitis (Gastrointestinal disorders) | 3
Dental Caries (Gastrointestinal disorders) | 2
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2
Hyperaesthesia Teeth (Gastrointestinal disorders) | 2
Lip Dry (Gastrointestinal disorders) | 1
Lip Oedema (Gastrointestinal disorders) | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 1
Tooth Fracture (Injury, poisoning and procedural complications) | 1
Migraine (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 1
Polycystic Ovaries (Reproductive system and breast disorders) | 1
Perioral Dermatitis (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
Anxiety (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/63/NCT04964063/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT04964063/SAP_001.pdf